CLINICAL TRIAL: NCT07329543
Title: Association of Advanced Glycation End-Product Burden With Response to Antiresorptive Therapy and Residual Fracture Risk in Osteoporosis: A Prospective Cohort Study
Brief Title: AGE Burden and Response to Antiresorptive Therapy in Osteoporosis
Status: Not yet recruiting | Type: Observational
Sponsor: Bursa City Hospital (Other Government)
Responsible Party: Principal Investigator, Taner Dandinoğlu, Principal Investigator, Bursa City Hospital
Other Study IDs: 2026-PMR-2
Record Dates: First submitted 2025-12-28; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Osteoporosis; Postmenopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis; Osteoporosis, Postmenopausal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Denosumab Group: Patients with osteoporosis receiving denosumab as part of routine clinical care.
- Bisphosphonate Group: Patients with osteoporosis receiving bisphosphonate therapy as part of routine clinical care.

SUMMARY:
Osteoporosis is a common condition that increases the risk of bone fractures. Although antiresorptive treatments such as bisphosphonates and denosumab are effective in increasing bone mineral density, some patients continue to experience fractures despite treatment.

Advanced glycation end-products (AGEs) accumulate in the body over time and can negatively affect bone quality by altering collagen structure and increasing inflammation. The role of AGE burden in predicting response to osteoporosis treatment has not been fully established.

This prospective cohort study aims to evaluate whether baseline AGE burden, measured non-invasively using skin autofluorescence, is associated with treatment response in patients receiving antiresorptive therapy for osteoporosis. Changes in bone mineral density, bone turnover markers, and fracture outcomes will be analyzed in relation to baseline AGE levels. The results of this study may help identify patients at risk for reduced treatment response and residual fracture risk.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years
* Diagnosis of osteoporosis based on dual-energy X-ray absorptiometry (DXA) criteria (T-score ≤ -2.5 at the lumbar spine, total hip, or femoral neck) or presence of a prior fragility fracture
* Planned initiation of antiresorptive therapy (denosumab or bisphosphonate) as part of routine clinical care
* Ability to undergo DXA measurements at baseline and during follow-up
* Ability and willingness to provide written informed consent

Exclusion Criteria:

* Diagnosis of diabetes mellitus (type 1 or type 2)
* Chronic kidney disease with estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m²
* Active malignancy or history of malignancy within the past 5 years
* Secondary causes of osteoporosis (including hyperparathyroidism, hyperthyroidism, Cushing's syndrome, malabsorption syndromes, or chronic liver disease)
* Use of medications known to significantly affect bone metabolism other than antiresorptive therapy (e.g., long-term systemic glucocorticoids, anabolic osteoporosis agents)
* Prior treatment with denosumab or bisphosphonates within the last 12 months
* Inflammatory rheumatic diseases or chronic inflammatory conditions that may affect bone metabolism
* Pregnancy or breastfeeding
* Inability to comply with study procedures or follow-up visits

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adults aged 50 years and older with a diagnosis of osteoporosis who are initiating antiresorptive therapy as part of routine clinical care. Participants will receive either denosumab or bisphosphonate treatment according to standard clinical indications. The study will prospectively evaluate the association between baseline advanced glycation end-product (AGE) burden and treatment response, including changes in bone mineral density, bone turnover markers, and fracture outcomes.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Percentage Change in Total Hip Bone Mineral Density | Baseline to 12 months
  Percentage change in total hip bone mineral density (BMD) from baseline to 12 months, measured by dual-energy X-ray absorptiometry (DXA), in relation to baseline advanced glycation end-product (AGE) burden.

SECONDARY OUTCOMES:
Percentage Change in Lumbar Spine Bone Mineral Density (L1-L4) | Baseline to 12 months
  Percentage change in lumbar spine (L1-L4) bone mineral density from baseline to 12 months measured by DXA.
Serum Concentration of Bone Turnover Markers (CTX and P1NP) | Baseline to 3 months and 12 months
  Changes in bone turnover markers, including serum C-terminal telopeptide of type I collagen (CTX) and procollagen type I N-terminal propeptide (P1NP), from baseline to 3 and 12 months.
Incident Fragility Fractures | Up to 12 months
  Occurrence of new fragility fractures during the follow-up period, assessed by patient report and medical records.
Association Between Baseline AGE Burden and Treatment Response | Baseline to 12 months
  Association between baseline AGE burden measured by skin autofluorescence and changes in bone mineral density and bone turnover markers during antiresorptive therapy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Sanguineti R, Puddu A, Mach F, Montecucco F, Viviani GL. Advanced glycation end products play adverse proinflammatory activities in osteoporosis. Mediators Inflamm. 2014;2014:975872. doi: 10.1155/2014/975872. Epub 2014 Mar 20. PMID 24771986